CLINICAL TRIAL: NCT01015131
Title: A Pilot Study to Evaluate the Correlation Between 18F-FLT-PET Uptake, Ki-67 Immunohistochemistry, and Proliferation Signature in Response to Neo-Adjuvant Chemotherapy in Breast Cancer
Brief Title: 18F-FLT-PET in Breast Cancer (MK-0000-139)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0000-139; 2009_692 (Other: Merck Registration Number)
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Results first posted 2012-12-20 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Participants (Experimental): 18F-FLT-PET imaging
  Interventions: Radiation: 18F-FLT-PET/CT Imaging

INTERVENTIONS:
Radiation: 18F-FLT-PET/CT Imaging — Participants receive the investigational radiotracer 18F-FLT intravenously and undergo Positron Emission Tomography (PET)/Computed Tomography (CT) scans at the following three times: prior to initiation of chemotherapy, at the end of the first cycle of treatment, and at the conclusion of chemotherapy.

SUMMARY:
This study correlated changes from baseline in Ki-67, an immunohistochemical marker of cell proliferation, with changes from baseline in tumor uptake of 3'-deoxy-3'[18F]-fluorothymidine (18F-FLT) following the first cycle of treatment with standard of care neo-adjuvant therapy in participants with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Has newly-diagnosed stage IIB/IIIA/IIIB locally advanced breast cancer
* Is eligible for pre-operative (neo-adjuvant) chemotherapy

Exclusion Criteria:

* Has a contraindication to magnetic resonance imaging (MRI)
* Any condition that would limit ability to undergo MRI or PET scans
* Is a nursing mother
* Has moderate to end-stage renal disease and is not on dialysis or has renal failure on chronic dialysis

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-04-08 (Actual); Primary Completion 2011-05-24 (Actual); Study Completion 2011-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After enrollment, 2 of the 46 participants discontinued due to lack of available 3'-deoxy-3'[18F]-fluorothymidine (18-FLT), leaving 44 participants as the baseline population.
Groups:
- All Participants: Participants who underwent 18-FLT positron emission tomography (PET) and standard of care (SOC) neo-adjuvant chemotherapy
Period: Overall Study
Arm/Group | All Participants
Started | 44
Completed | 36
Not Completed | 8
Not completed — Physician Decision | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 2
Not completed — Other Protocol Specified Criteria | 4

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 18F-FLT-PET Mean Standardized Uptake Value (SUVmean) After the First Cycle of Standard of Care (SOC) Neo-adjuvant Chemotherapy.
Description: Participants undergo a baseline 18F-FLT-PET/CT scan followed by a magnetic resonance imaging (MRI) scan prior to chemotherapy. These scans are repeated in approximately 2 to 3 weeks, at the end of the first cycle of chemotherapy to derive a standardized uptake value (SUV) of 18F-FLT, which is calculated from the ratio of radioactivity concentration within a region of interest, and the injected dose at the time of injection, divided by body weight. The SUVmean averages the radioactivity values within a region of interest.
Time Frame: Baseline and up to 3 weeks
Population: Participants whose SUV were measured at Baseline and after 1 cycle of chemotherapy
Measure: Mean (Standard Deviation); unit: SUV
Arm/Group | All Participants
Number analyzed (Participants) | 36
SUV
  Baseline | 2.79 (1.36)
  End of Cycle 1 | 1.78 (1.03)
  Change from Baseline | 1.00 (0.95)

2. Secondary Outcome: Change From Baseline in Proliferation Signature Score (PSS) After the First Cycle of SOC Neo-adjuvant Chemotherapy.
Description: Core needle biopsies (CNBs) obtained at baseline and after approximately 2-3 weeks of treatment, at the end of the first cycle of chemotherapy, are used to measure cell proliferation by a Proliferation Signature Score (PSS). PSS is calculated from the messenger RNA (mRNA) expression of 47 genes that negatively correlate with time to recurrence, and involves taking their average normalized scores. For reference, a database of 16,000 tumors gave a minimum PSS of 1.51 and a maximum PSS of 2.89; where a higher PSS is associated with an increase in proliferation, higher tumor grade and worse outcomes.
Time Frame: Baseline and up to 3 weeks
Population: Participants who had PSS determined at Baseline and after 1 cycle of chemotherapy
Measure: Mean (Standard Deviation); unit: Proliferation Score
Arm/Group | All Participants
Number analyzed (Participants) | 35
Proliferation Score
  Baseline (n = 36) | 2.34 (0.13)
  End of Cycle 1 | 2.20 (0.21)
  Change from Baseline | 0.15 (0.21)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority or Other; p < 0.01, paired t-test; Mean Difference (Final Values) = 0.1521, 90% CI 2-sided [0.0932 to 0.2111]

3. Secondary Outcome: Change From Baseline in Tumor Volume at the End of SOC Neo-adjuvant Chemotherapy.
Description: MRI of participants was used to measure tumor volumes at baseline and after completing chemotherapy, after approximately 11 to 30 weeks of treatment.
Time Frame: Baseline and up to 30 weeks
Population: Participants who had tumors measured by MRI at Baseline and at the end of chemotherapy
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | All Participants
Number analyzed (Participants) | 36
cm^3
  Baseline | 22.74 (30.82)
  End of Chemotherapy | 6.14 (14.69)
  Change from Baseline | 16.59 (29.57)

4. Secondary Outcome: Spearman's Rank Correlation Coefficient Between Change From Baseline in PSS After the First Cycle of SOC Neo-adjuvant Chemotherapy, and Change From Baseline in Tumor Volume at the End of SOC Neo-adjuvant Chemotherapy.
Description: The Spearman's rank correlation coefficient was computed by ranking the data and using the ranks in the Pearson product-moment correlation formula. In case of ties, the averaged ranks were used.
Time Frame: Baseline and up to 30 weeks
Population: Participants who had their PSS measured after 1 cycle of chemotherapy and their tumors measured at the end of chemotherapy
Measure: Number (90% Confidence Interval); unit: Correlation coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 35
Correlation coefficient | 0.20 (0.21) [-0.09 to 0.45]

5. Secondary Outcome: Spearman's Rank Correlation Coefficient Between Change From Baseline in Ki-67 LI After the First Cycle of SOC Neo-adjuvant Chemotherapy, and Change From Baseline in Tumor Volume at the End of SOC Neo-adjuvant Chemotherapy.
Description: as for outcome 4
Time Frame: Baseline and up to 30 weeks
Population: Participants who had their Ki-67 LI measured after 1 cycle of chemotherapy and their tumors measured at the end of chemotherapy
Measure: Number (90% Confidence Interval); unit: Correlation coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 32
Correlation coefficient | 0.13 [-0.18 to 0.41]

6. Primary Outcome: Change From Baseline in 18F-FLT-PET Maximum Standardized Uptake Value (SUVmax) After the First Cycle of SOC Neo-adjuvant Chemotherapy.
Description: Participants undergo a baseline 18F-FLT-PET/CT scan followed by a magnetic resonance imaging (MRI) scan prior to chemotherapy. These scans are repeated in approximately 2 to 3 weeks, at the end of the first cycle of chemotherapy to derive a standardized uptake value (SUV) of 18F-FLT, which is calculated from the ratio of tissue radioactivity concentration within a region of interest, and the injected dose at the time of injection, divided by body weight. The SUVmax measures the maximum radioactivity values within a region of interest.
Time Frame: Baseline and up to 3 weeks
Population: Participants whose SUV were measured at Baseline and after 1 cycle of chemotherapy
Measure: Mean (Standard Deviation); unit: SUV
Arm/Group | All Participants
Number analyzed (Participants) | 36
SUV
  Baseline | 5.76 (2.83)
  End of Cycle 1 | 3.52 (2.13)
  Change from Baseline | 2.24 (1.99)

7. Primary Outcome: Change From Baseline in Ki-67 Labeling Index After the First Cycle of SOC Neo-adjuvant Chemotherapy.
Description: Core needle biopsies (CNB) are obtained after completing imaging studies at baseline and approximately 2 to 3 weeks later, after the first cycle of chemotherapy. These tissue samples are then used to measure expression of the cell proliferation marker Ki-67, by manually counting percentage positive immunostained cells, denoted the labeling index (LI).
Time Frame: Baseline and up to 3 weeks
Population: Participants whose Ki-67 Labeling Index were measured at Baseline and after 1 cycle of chemotherapy
Measure: Mean (Standard Deviation); unit: Labeling Index
Arm/Group | All Participants
Number analyzed (Participants) | 32
Labeling Index
  Baseline (n = 36) | 57.89 (28.17)
  End of Cycle 1 | 43.81 (31.80)
  Change from Baseline | 10.53 (20.64)

8. Primary Outcome: Spearman's Rank Correlation Coefficient Between Change From Baseline in Ki-67 Labeling Index and Change From Baseline in SUVmean After the First Cycle of SOC Neo-adjuvant Chemotherapy.
Description: as for outcome 4
Time Frame: Baseline and up to 3 weeks
Population: Participants who had both their changes from baseline in Ki-67 LI and SUVmean determined at the end of Cycle 1 of chemotherapy.
Measure: Number (90% Confidence Interval); unit: Correlation coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 32
Correlation coefficient | 0.53 [0.28 to 0.72]

9. Primary Outcome: Spearman's Rank Correlation Coefficient Between Change From Baseline in Ki-67 Labeling Index and Change From Baseline in SUVmax After the First Cycle of SOC Neo-adjuvant Chemotherapy.
Description: as for outcome 4
Time Frame: Baseline and up to 3 weeks
Population: Participants who had both their changes from baseline in Ki-67 LI and SUVmax determined at the end of Cycle 1 of chemotherapy.
Measure: Number (90% Confidence Interval); unit: Correlation coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 32
Correlation coefficient | 0.46 [0.19 to 0.67]

10. Secondary Outcome: Spearman's Rank Correlation Coefficient Between Change From Baseline in SUVmax After the First Cycle of SOC Neo-adjuvant Chemotherapy, and Change From Baseline in Tumor Volume at the End of SOC Neo-adjuvant Chemotherapy.
Description: as for outcome 4
Time Frame: Baseline and up to 30 weeks
Population: Participants who had their SUVmax measured after 1 cycle of chemotherapy and their tumors measured at the end of chemotherapy
Measure: Number (90% Confidence Interval); unit: Correlation coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 36
Correlation coefficient | 0.22 [-0.06 to 0.47]

11. Secondary Outcome: Spearman's Rank Correlation Coefficient Between Change From Baseline in SUVmean After the First Cycle of SOC Neo-adjuvant Chemotherapy, and Change From Baseline in Tumor Volume at the End of SOC Neo-adjuvant Chemotherapy.
Description: as for outcome 4
Time Frame: Baseline and up to 30 weeks
Population: Participants who had their SUVmean measured after 1 cycle of chemotherapy and their tumors measured at the end of chemotherapy
Measure: Number (90% Confidence Interval); unit: Correlation coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 36
Correlation coefficient | 0.20 [-0.08 to 0.45]

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 8/44
Other Adverse Events (participants affected / at risk) | 39/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=44)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (5)
Rectal bleeding (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=44)
Anaemia (Blood and lymphatic system disorders) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 17 (34)
Constipation (Gastrointestinal disorders) | 9 (10)
Diarrhoea (Gastrointestinal disorders) | 4 (6)
Haemorrhoids (Gastrointestinal disorders) | 3 (3)
Heartburn (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 23 (33)
Stomatitis (Gastrointestinal disorders) | 5 (14)
Fatigue (General disorders) | 8 (8)
Fever (General disorders) | 4 (6)
Mucositis (General disorders) | 8 (10)
Oedema (General disorders) | 3 (3)
Weakness generalised (General disorders) | 3 (3)
Hypersensitivity reaction (Immune system disorders) | 3 (3)
Common cold (Infections and infestations) | 3 (5)
Incision site pain (Injury, poisoning and procedural complications) | 8 (8)
Alanine aminotransferase increased (Investigations) | 3 (3)
Haemoglobin decreased (Investigations) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 8 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (14)
Dizziness (Nervous system disorders) | 5 (5)
Headache (Nervous system disorders) | 5 (5)
Neuropathy (Nervous system disorders) | 6 (6)
Insomnia (Psychiatric disorders) | 6 (6)
Breast pain (Reproductive system and breast disorders) | 3 (3)
Postmenopausal symptoms (Reproductive system and breast disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4)
Nail changes (Skin and subcutaneous tissue disorders) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.